CLINICAL TRIAL: NCT02621450
Title: The Effect of Low Sodium Dialysate on Ambulatory Blood Pressure Measurement Parameters in Patients Undergoing Hemodialysis
Brief Title: Low Sodium Dialysate and Ambulatory Blood Pressure Measurement Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hasan ali gümrükçüoğlu, associated professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2012-51
Record Dates: First submitted 2015-11-21; First posted 2015-12-03 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Renal Failure; Hypertension
Keywords: chronic renal failure; hypertension; ampulatory blood pressure
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standart dialysate (Placebo Comparator): dialysate sodium 140 mEq/L
  Interventions: Biological: standart dialysis
- low sodium dialysate (Other): dialysate sodium will be reduced from 140 mEq/L to 137 mEq/L
  Interventions: Biological: low sodium dialysis

INTERVENTIONS:
Biological: standart dialysis — dialysate sodium consentration 140 mEq
  Arms: standart dialysate
Biological: low sodium dialysis — dialysate sodium consentration will be reducer from 140 mEq to 137 mEq
  Arms: low sodium dialysate

SUMMARY:
End stage renal disease (ESRD) is related with increased cardiovascular mortality and morbidity. Hypertension (HT) is an important risk factor for cardiovascular disorder among hemodialysis (HD) patients. The aim of this study going to investigate the effectivity of low-sodium dialysate on the systolic and diastolic blood pressure (BP) levels detected by ABPM and interdialytic weight gain (IDWG) in patients undergoing sustained hemodialysis treatment.

Methods: The study will be included 46 patients who had creatinine clearance levels less than 10 ml/min/1.73 m2 and had been on chronic HD treatment for at least one year. After the enrollment stage, the patients will be allocated low-sodium dialysate or standard-sodium dialysate for six months via computer-generated randomization.

DETAILED DESCRIPTION:
Patient Selection The present study is a single-center, randomized controlled and double blinded trial. The patients going to enroll for this study had creatinine clearance less than 10 ml/min/1.73 m2 and had been on intermittent HD treatment for at least one year.

The exclusion criteria for the present study are masking or white coat hypertension, heart failure, cardiomyopathies, acute coronary syndromes, chronic ischemic heart disease, acute or chronic liver disease, endocrine or pulmonary diseases, valvular heart diseases, malignancies, active urinary tract infections, hemoglobin levels below 8 g/dL, and hypotension tendency.

Sixty-four patients going to enroll for eligibility and after the initial assessment. Clinic and laboratory profiles of the patients including cause of renal disease, history of HT and antihypertensive treatments going to record by systematic review of the patient files. After the enrollment stage, the patients going to allocate low-sodium dialysate or standard sodium dialysate for 6 months via computer-generated randomization.

They going to dialyze three times a week with synthetic polysulfone (Hollow-fiber, Low Flux, KUF<20, 1.6 m2) membrane, each session lasting 4 hours with bicarbonate dialysate (with 33mmol/L concentration) and 300-350 ml/min blood-flow. .

Study protocol All patients going to assess before and 6 months after the study. Before initiating the study, all patients were dialyzed with 140 mEq/L sodium concentration. In the low-sodium dialysate group, the dialysate sodium concentration going to reduce from 140 to 137mEq/L. To eliminate the acute effects of hemodialysis on the parameters measured, baseline and end-of-study measurements going to perform in non-dialysis day, 24 hours after the mid-week session.

Ambulatory blood pressure measurement Ambulatory BP measurement during 24-hour going to perform using a Space Labs 90207 oscillometric method (Redmond, Washington, USA). The BP measurements going to perform automatically from non-fistula arm. The confirmation of the device going to check with the standard auscultator method in order to ensure that the changes in BP values between the two methods did not exceed +5 mm Hg.

The device going to set to achieve BP evaluation at 30-minute intervals during the night (11:00 PM to 07:00 AM) and at 20-minute intervals during the day (07:00 AM to 11:00 PM).

''Nocturnal dipping'' going to define as a decrease of greater than 10% (when compared with the daytime values) in the systolic or diastolic blood pressure at night. ''Non-nocturnal dipping'' going to define as a decrease of less than 10% (when compared with the daytime values) in the blood pressure parameters levels at night or did not decrease in the systolic or diastolic blood pressure at night

ELIGIBILITY:
Inclusion Criteria:

The patients with creatinine clearance less than 10 ml/min/1.73 m2 and under intermittent HD treatment for at least one year are included into the study.

Exclusion Criteria as follows:

Masking or white coat hypertension, heart failure, cardiomyopathies, acute coronary syndromes, chronic ischemic heart disease, acute or chronic liver disease, endocrine or pulmonary diseases, valvular heart diseases, malignancies, active urinary tract infections, hemoglobin levels below 8 g/dL, and hypotension tendency -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure measurement | six months

CONTACTS AND LOCATIONS:
Overall Officials: hasan ali gümrükçüoğlu, Principal Investigator — Yuzuncu Yil Univesty

REFERENCES:
- [Background] Gumrukcuoglu HA, Ari E, Akyol A, Akdag S, Simsek H, Sahin M, Gunes Y, Tuncer M. Effects of lowering dialysate sodium on carotid artery atherosclerosis and endothelial dysfunction in maintenance hemodialysis patients. Int Urol Nephrol. 2012 Dec;44(6):1833-9. doi: 10.1007/s11255-011-0117-5. Epub 2012 Jan 14. PMID 22246593
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822